CLINICAL TRIAL: NCT03464513
Title: Role of MSCT Angiography in Evaluation of Lower Gastrointestinal Bleeding
Brief Title: MSCT Angiography in Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Gergis Naeem, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Angiography
Record Dates: First submitted 2018-02-23; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Lower Gastrointestinal Bleeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with GIT bleeding (Other): Patients with active lower Gastrointestinal bleeding
  Interventions: Device: Multislice CT Angiography

INTERVENTIONS:
Device: Multislice CT Angiography — Multislice CT angiography (MSCTA) provides a relatively non-invasive and effective way of localising the source of bleeding, especially in patients with continuous bleeding.

SUMMARY:
Lower gastrointestinal bleeding occurs distal to the ligament of treitz and may involve the small bowel, colon and rectum .

Active lower gastrointestinal bleeding is a common, potentially life threatening medical presentation that can be challenging to localize and treat .

There are many diseases that may cause lower gastrointestinal bleeding, including angiodysplasia, diverticulosis, benign or malignant bowel neoplasm, inflammatory bowel disease, ischemic bowel disease, and infectious bowel disease.

Often, gastrointestinal bleeding will stop spontaneously, but in approximately 25% of patients, bleeding is massive or recurrent, requiring imaging localization and directed therapy.

DETAILED DESCRIPTION:
Accurate and prompt diagnosis of the bleeding source is crucial because mortality can be as high as 40%if there is hemodynamic instability in patients .

Because of the length of GI tract, the multitude of pathologic processes that can result in GI bleeding, imaging plays a primary role in the diagnosis .

Multislice CT angiography (MSCTA) provides a relatively non-invasive and effective way of localising the source of bleeding, especially in patients with continuous bleeding .

MSCTA is being increasingly used because it is a widely available, non-invasive and fast diagnostic technique that allows for the visualization of the entire intestinal tract and its lesions, the identification of the vascularity and possible vascular abnormalities. In addition, this technique does not require preparation in patients with acute bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to assiut university hospital with active lower gastrointestinal bleeding.

Exclusion Criteria:

* Patients whom are sensitive to contrast. Pregnant women. Patients with renal insufficiency

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
MSCTA in the evaluation of patients presenting with active lower gastrointestinal bleeding. | 1 hour
  Multislice ct angiography

REFERENCES:
- [Background] Yoon W, Jeong YY, Shin SS, Lim HS, Song SG, Jang NG, Kim JK, Kang HK. Acute massive gastrointestinal bleeding: detection and localization with arterial phase multi-detector row helical CT. Radiology. 2006 Apr;239(1):160-7. doi: 10.1148/radiol.2383050175. Epub 2006 Feb 16. PMID 16484350